CLINICAL TRIAL: NCT04860219
Title: The Prospect of Lactoferrin Use as Adjunctive Agent in Management of SARS COV-2 Patients: A Randomized Pilot Study
Brief Title: Lactoferrin Use in (SARS-CoV-2) Management
Acronym: SARS-CoV-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mohamed E Ghoniem, Associate Professor of Internal Medicine- Faculty of Medicine, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-1937
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Lactoferrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): None of the participants in the Control Group received lactoferrin
- 200 mg lactoferrin orally once daily Group (Active Comparator): received 200 mg lactoferrin orally once daily
  Interventions: Dietary Supplement: Lactoferrin
- 200 mg lactoferrin orally twice daily Group (Active Comparator): received 200 mg lactoferrin orally twice daily
  Interventions: Dietary Supplement: Lactoferrin

INTERVENTIONS:
Dietary Supplement: Lactoferrin — 7 successive days treatment of Lactoferrin started within day 0 of COVID-19 diagnosis by RT-PCR
  Arms: 200 mg lactoferrin orally once daily Group; 200 mg lactoferrin orally twice daily Group

SUMMARY:
Background: Preventive, adjunctive and curative properties of lactoferrin have been evaluated since the first wave of severe acute respiratory syndrome coronavirus (SARS-CoV), viral respiratory disease, emerged 18 years ago. Despite the discovery of new vaccine candidates, there is currently no widely approved treatment for SARS-CoV-2 (COVID-19). Strict adherence to infection prevention and control procedures, as well as vaccines, can, however, prevent the spread of SARS-CoV-2. Objective: Hence, this study evaluated the efficacy of lactoferrin treatment in improving clinical symptoms and laboratory indices among individuals with mild to moderate coronavirus disease-19 (COVID-19). Design and Participants: A randomized, prospective, interventional pilot study conducted between July 8 and September 18, 2020 used a hospital-based sample of 54 laboratory confirmed participants with mild to moderate symptoms of COVID-19. Randomization into a control and two treatment groups ensured all groups received the approved Egyptian COVID-19 management protocol; only treatment group participants received lactoferrin at different doses for seven days. Clinical symptoms and laboratory indices were assessed on Days 0, 2 and 7 after starting treatments. Mean values with standard deviation and one-way analysis of variance with least significant difference post hoc of demographic and laboratory data between control and treatment groups were calculated. Key Results: Our study showed no stastically significant difference among studied groups regarding recovery of symptoms or laboratory improvement. Conclusion: Further research into therapeutic properties particularly related to dosage, duration and follow-up after treatment with lactoferrin in individuals with COVID-19 is required.

ELIGIBILITY:
Inclusion Criteria:

1. participants over 20 years of age
2. positive for nasopharyngeal swab reverse transcriptase polymerase chain reaction (RT-PCR) for COVID-19
3. blood oxygen saturation (SpO2) > 93%.

Exclusion criteria:

1. pregnant and breastfeeding women
2. individuals confirmed to be allergic to milk protein
3. those with a medical history of bronchial hyperactivity or pre-existing respiratory diseases
4. ICU inpatients with COVID-19.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
time to be symptoms free and normal laboratory results | 7 days after enrollment
  duration from day 0 symptoms till 7 days symptoms free and normal laboratory findings

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine -Zagazig University, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
The datasets generated and/or analyzed during the current study are available from the corresponding author upon request.